CLINICAL TRIAL: NCT04152486
Title: Evaluation of a Heterologous, Two-dose Preventive Ebola Vaccine for Effectiveness and Safety in the Democratic Republic of the Congo
Brief Title: Effectiveness and Safety of a Heterologous, Two-dose Ebola Vaccine in the DRC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Epicentre (Other); Ministère de la Santé de la RDC (Unknown); Médecins Sans Frontières, France (Other); Coalition for Epidemic Preparedness Innovations (Other); Janssen Vaccines & Prevention B.V. (Industry); Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DRC-EB-001
Record Dates: First submitted 2019-10-25; First posted 2019-11-05 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-06

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Intervention Model Description: Single arm, open-label, non-randomized interventional trial of the two dose, Ad26.ZEBOV, MVA-BN-Filo Ebola preventative vaccine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): The vaccine Ad26.ZEBOV (5x10^10 viral particles (vp)) will be given as the first dose and the vaccine MVA-BN-Filo (1x10^8 infectious units (Inf U)) will be given as the second dose 56 (-14 day +28 day) days later.
  Interventions: Biological: Ad26.ZEBOV, MVA-BN-Filo vaccine

INTERVENTIONS:
Biological: Ad26.ZEBOV, MVA-BN-Filo vaccine — Ad26.ZEBOV: a monovalent vaccine expressing the full-length glycoprotein (GP) from Ebola virus (EBOV) Mayinga. The vaccine is produced in the human cell line PER.C6®.
  MVA-mBN226B: further referred to as Modified Vaccinia Ankara (MVA)-BN®-Filo. This is a multivalent vaccine expressing the EBOV GP, the Sudan virus (SUDV) GP, the Marburg virus (MARV) Musoke GP, and the Taï Forest virus (TAFV, formerly known as Côte d'Ivoire ebolavirus) nucleoprotein (NP). The EBOV GP expressed by MVA BN Filo has 100% homology with the one expressed by Ad26.ZEBOV.

SUMMARY:
A single arm, open-label, non-randomized, interventional phase 3 study to measure safety and effectiveness of a heterologous, two dose preventative vaccine (Ad26. ZEBOV, MVA-BN®-Filo) against Ebola Virus Disease.

DETAILED DESCRIPTION:
Ebola Virus Disease (EVD) is an acute, systemic, febrile syndrome caused by Ebola viruses. EVD has a case fatality ranging from 30% to 90% and spreads by direct contact with body fluids of symptomatic patients.

During the 2013-16 Ebola outbreak in Guinea, a Phase 3 cluster-randomised ring-vaccination trial using single-dose rVSV-ZEBOV-GP investigational vaccine reported 100% efficacy in protection against EVD. In 2016, the WHO Strategic Advisory Group of Experts (SAGE) on Immunization recommended the rapid deployment of rVSV-ZEBOV-GP in case of an EVD outbreak under an Expanded Access (compassionate use) protocol, with informed consent and Good Clinical Practice (GCP) compliance.

A new EVD outbreak started in North Kivu and Ituri provinces in the Democratic Republic of Congo in July 2018. Despite extensive control measures, including vaccination with rVSV-ZEBOV-GP in active outbreak areas, the outbreak has continued and WHO declared the outbreak a Public Health Emergency of International Concern on 17 July 2019. The ongoing outbreak has prompted consideration of additional vaccine candidates that might assist in preventing the spread of this infection to currently unaffected communities.

This study will investigate population-level vaccination with a two-dose prophylactic vaccine against Ebola, the Ad26.ZEBOV, MVA-BN-Filo vaccine that has been extensively studied in 11 previous safety and immunogenicity trials. This will be done by offering vaccination first to communities that neighbour the outbreak area or that are located on transport routes from the edge of the outbreak area to major centres like Goma.

In this study, approximately 500,000 healthy adults and children will be given the two-dose candidate vaccine regimen VAC52150 that consists of two vaccines, Ad26.ZEBOV and MVA-BN®-Filo, administered at an interval of 56 days (-14 day +28 day). Safety will be assessed in a safety subset of 1000 individuals and a pregnancy subset of up to 500 pregnant women will be followed to delivery. The first 100 infants born to these pregnant participants will be given a clinical examination at 3 months post-delivery. The study will estimate vaccine coverage of dose 1 and dose 2 overall and in different target groups and will also examine the knowledge and perceptions of persons eligible for large-scale delivery of a preventative Ebola vaccine with a two-dose vaccine strategy. The effectiveness of the vaccination on EVD will be determined through a test-negative case control study. The target sample size for the primary effectiveness evaluation is 110 laboratory-confirmed EVD cases.

An exploratory objective is to assess the immune response at before the second dose and 21 days after the second dose (MVN-BN-Filo) in a subgroup of 50 adults and 50 children who receive dose 2 beyond the recommended 56-day interval.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide a written or witnessed (if illiterate) informed consent form indicating that he or she understands the reasons for the study and is willing to participate in the study and be vaccinated. If less than 18 years old, must have a parent or guardian that is able to meet this criterion.
2. Must be aged 1 year or older.
3. Must be healthy in the investigator's clinical judgment as assessed on the day of vaccination.
4. Must be willing to have a photograph taken.
5. Participant must be available and willing to participate for duration of study visits and follow up.

Exclusion Criteria:

1. Known history of Ebola virus disease.
2. Has received any experimental Ebola vaccine less than one month prior to Visit 1.
3. Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products, egg and egg proteins or gentamicin.
4. Presence of acute illness (excluding minor illnesses such as mild diarrhea or mild upper respiratory tract infection) or temperature ≥38.0ºC at Visit 1 (dose 1 visit). Participants with such symptoms will be temporarily excluded from vaccination at that time but may be rescheduled for vaccination at a later date if feasible.
5. Presence of significant conditions or clinically significant findings at the vaccination visit for which, in the opinion of the investigator, vaccination would not be in the best interest of the participant.
6. History of recurrent generalized hives.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20426 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Numbers and odds of vaccination status in Ebola Virus Diseases cases and in EVD-negative controls. | Through study completion, an average of 2 years.
  Test negative case control study of 110 laboratory confirmed EVD cases matched to controls who test negative for EVD. Effectiveness is derived from the odds ratio for vaccination in cases compared to controls to calculate vaccine effectiveness.

SECONDARY OUTCOMES:
Number and proportion of adults and children with solicited and unsolicited serious adverse events. | From date of first vaccination to the one month post-dose 2 assessment of the last vaccinated participant.
  Data on SAEs within one month post-dose 2 that are considered related to vaccination with Ad26. ZEBOV, MVA-BN®-Filo vaccine in adults and children.
Number and proportion of adults and children receiving dose 1. | From date of first vaccination up to month 12.
  Vaccine uptake
Number and proportion of adults and children receiving dose 2. | From date of first vaccination up to month 12.
  Vaccine coverage
Number of participants participating in in-depth interviews and focus group discussions | Through to study completion at month 24.
  Focus group discussions and in-depth interviews on participant and community perceptions of the trial and on vaccine acceptability.

OTHER OUTCOMES:
Samples collected for immunogenicity subset at 2 time points | From date of dose 2 through to 21 days post-dose 2.
  Level of immunoglobulin G binding antibodies at dose 2 and 21 days post-dose 2

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Muyembe-Tamfum, MD, PhD, Principal Investigator — L'Institut National de Recherche Biomédicale RDC; Daniel Bausch, MD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Deborah Watson-Jones, MD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- L'Institut National de Recherche Biomédicale RDC, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
Individual level data (de-identified) that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Six months to 60 months after publication of main trial results.
Access Criteria: Access request to:
  Deborah.Watson-Jones@lshtm.ac.uk (ORCID: 0000-0001-6247-1746) cc. Tansy Edwards@lshtm.ac.uk (ORCID: 0000-0002-6110-014X) cc. Edward.Choi@lshtm.ac.uk (ORCID: 0000-0002-8148-120X)

REFERENCES:
- [Derived] Watson-Jones D, Kavunga-Membo H, Grais RF, Ahuka S, Roberts N, Edmunds WJ, Choi EM, Roberts CH, Edwards T, Camacho A, Lees S, Leyssen M, Spiessens B, Luhn K, Douoguih M, Hatchett R, Bausch DG, Muyembe JJ; DRC-EB-001 protocol writing team. Protocol for a phase 3 trial to evaluate the effectiveness and safety of a heterologous, two-dose vaccine for Ebola virus disease in the Democratic Republic of the Congo. BMJ Open. 2022 Mar 8;12(3):e055596. doi: 10.1136/bmjopen-2021-055596. PMID 35260458